CLINICAL TRIAL: NCT05137067
Title: Effectiveness of RaproCell in Alleviating the Side Effects of Chemotherapeutic Agents, Without Adversely Impacting the Overall Success of the Agents on Cancer Cells.
Brief Title: A Novel Approach for Alleviating the Side Effects of Chemotherapeutic Agents.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Optimal Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPC006
Record Dates: First submitted 2021-04-11; First posted 2021-11-30 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Lung Cancer; Prostate Cancer
Keywords: Cancer Breast Lung Prostate
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized interventional parallel study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active product and placebo will be in identical packets.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Chemotherapeutic agent A (Docetaxel) (Other): The patients with breast cancer will receive chemotherapeutic agent A
  Interventions: Drug: Chemotherapeutic agent A(Docetaxel),B(Cisplatin) or C(Docetaxel).
- Chemotherapeutic agent A (Docetaxel) plus placebo (Placebo Comparator): The patients with breast cancer will receive chemotherapeutic agent A plus a placebo.
  Interventions: Drug: Chemotherapeutic agent A(Docetaxel),B(Cisplatin) or C(Docetaxel) plus placebo
- Chemotherapeutic agent A (Docetaxel) plus RaproCell (Active Comparator): The patients with breast cancer will receive chemotherapeutic agent A plus RaproCell.
  Interventions: Dietary Supplement: Chemotherapeutic agent A(Docetaxel),B(Cisplatin) or C(Docetaxel) plus Dietary Supplement (RaproCell)
- Chemotherapeutic agent B (Cisplatin) (Other): The patients with lung cancer will receive Chemotherapeutic agent B
  Interventions: Drug: Chemotherapeutic agent A(Docetaxel),B(Cisplatin) or C(Docetaxel).
- Chemotherapeutic agent B (Cisplatin) plus placebo (Placebo Comparator): The patients with lung cancer will receive Chemotherapeutic agent B plus placebo.
  Interventions: Drug: Chemotherapeutic agent A(Docetaxel),B(Cisplatin) or C(Docetaxel) plus placebo
- Chemotherapeutic agent B (Cisplatin) plus RaproCell (Active Comparator): The patients with lung cancer will receive Chemotherapeutic agent B plus RaproCell.
  Interventions: Dietary Supplement: Chemotherapeutic agent A(Docetaxel),B(Cisplatin) or C(Docetaxel) plus Dietary Supplement (RaproCell)
- Chemotherapeutic agent C (Docetaxel) (Other): The patients with prostate cancer will receive Chemotherapeutic agent C
  Interventions: Drug: Chemotherapeutic agent A(Docetaxel),B(Cisplatin) or C(Docetaxel).
- Chemotherapeutic agent C (Docetaxel) plus placebo (Placebo Comparator): The patients with prostate cancer will receive Chemotherapeutic agent C plus placebo.
  Interventions: Drug: Chemotherapeutic agent A(Docetaxel),B(Cisplatin) or C(Docetaxel) plus placebo
- Chemotherapeutic agent C plus (Docetaxel) RaproCell (Active Comparator): The patients with prostate cancer will receive Chemotherapeutic agent C plus RaproCell.
  Interventions: Dietary Supplement: Chemotherapeutic agent A(Docetaxel),B(Cisplatin) or C(Docetaxel) plus Dietary Supplement (RaproCell)

INTERVENTIONS:
Dietary Supplement: Chemotherapeutic agent A(Docetaxel),B(Cisplatin) or C(Docetaxel) plus Dietary Supplement (RaproCell) — Chemotherapeutic side effect elimination without adversely effecting the Chemotherapeutic agent drug.
  Other Names: RaproCell
  Arms: Chemotherapeutic agent A (Docetaxel) plus RaproCell; Chemotherapeutic agent B (Cisplatin) plus RaproCell; Chemotherapeutic agent C plus (Docetaxel) RaproCell
Drug: Chemotherapeutic agent A(Docetaxel),B(Cisplatin) or C(Docetaxel) plus placebo — Placebo
  Arms: Chemotherapeutic agent A (Docetaxel) plus placebo; Chemotherapeutic agent B (Cisplatin) plus placebo; Chemotherapeutic agent C (Docetaxel) plus placebo
Drug: Chemotherapeutic agent A(Docetaxel),B(Cisplatin) or C(Docetaxel). — Chemotherapeutic agent A(Docetaxel),B(Cisplatin) or C(Docetaxel).
  Arms: Chemotherapeutic agent A (Docetaxel); Chemotherapeutic agent B (Cisplatin); Chemotherapeutic agent C (Docetaxel)

SUMMARY:
This study will assess the effectiveness of a natural nutraceutical in treating the known side effects of chemotherapeutic agents in cancer patients.

DETAILED DESCRIPTION:
This study will assess the effectiveness of a natural nutraceutical in treating the known side effects of chemotherapeutic agents in cancer patients. The study will be observing the standard treatment protocol for any degradation or enhancement due to the nutraceutical.

ELIGIBILITY:
Inclusion Criteria:

Active breast cancer patients taking one of the studies listed drugs within the age range.

Active lung cancer patients taking one of the studies listed drugs within the age range.

Active prostate cancer patients taking one of the studies listed drugs within the age range.

-

Exclusion Criteria:

Anyone without the three types of cancer (breast cancer, lung cancer, prostate cancer) listed in inclusion criteria.

-

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer: Female only
  Lung cancer: Both Female and Male
  Prostate cancer: Male
Enrollment: 90 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
PROMIS (Patient-Reported Outcomes Measurement Information System) Global 10 Health Questionnaire to assess change from baseline. | Once a week for 3 months
  A summary indicator of health status by assessing 5 domains: physical function, fatigue, pain, emotional distress, and social health to assess change from baseline for improvement or decline.
Symptom Assessment Questionnaire to assess change from baseline. | Once a week for 3 months
  A symptom is a sensation or perception of change related to health function experienced by an individual. Symptoms such as fatigue, pain and nausea can be classified according to their severity and perceived impact on function as a change from baseline for improvement or decline.

SECONDARY OUTCOMES:
Cancer antigens blood markers to assess change from baseline. | Once a week for 3 months.
  Breast: CA 27.29, serial monitor report; carcinoembryonic antigen (CEA), serial monitor report; lipid-associated sialic acid (LASA), serial monitor report. Lung: Carcinoembryonic antigen (CEA), serial monitor report; lipid-associated sialic acid (LASA), serial monitor report; neuron-specific enolase (NSE), serial monitor report. Prostate: Prostate-specific antigen (PSA), serial monitor report; prostatic acid phosphatase (PAP), serial monitor report as a change from baseline for improvement or decline.

CONTACTS AND LOCATIONS:
Overall Officials: EA Jeppsen, MD, Study Chair — Optimal Health Clinic; Steven Osguthorpe, ND, Principal Investigator — Optimal Health Research
Locations (1):
- Optimal Health Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No